CLINICAL TRIAL: NCT04477135
Title: Investigation of the Relationship Between Upper Extremity Pain and Ultrasound Use in Perinatologist
Brief Title: Upper Extremity paın and Ultrasound Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nefise Nazlı YENIGUL (Other)
Responsible Party: Sponsor-Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Organization: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20.11.29
Record Dates: First submitted 2020-07-03; First posted 2020-07-20 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Pain, Chronic; Upper Extremity Problem
MeSH Terms: conditions — Chronic Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- perinatologists (Other): perinatologists working actively and performing ultrasonography every day
  Interventions: Other: upper extremity pain; Procedure: ultrasonography

INTERVENTIONS:
Other: upper extremity pain — upper extremity pain in perinatologists due to working actively and performing ultrasonography every day
Procedure: ultrasonography — ultrasonography

SUMMARY:
The relationship between perinatologists' ultrasound use and upper limb joint pain will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Those who have received specialization training in the branch of perinatology and have completed their specialty in the branch and worked as a perinatologist
* Those who want to participate in the study

Exclusion Criteria:

* Patients with discomfort and operation in the upper limb prior to perinatology training
* Physicians in other branches

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Upper extremity pain in perinatologists | 2 month
  The relationship between perinatologists' ultrasound use and upper extremity pain. Perinatologists use ultrasound for a long time during the day. This can cause some pain in the upper extremities. In our study, the investigators will have a survey of perinatologists and ask some questions: How long have they been doing this profession, which hands they use, how many patients they examine per day, do they have any complaints of upper extremity. The investigators will try to relate upper extremity pain with their answers.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided